CLINICAL TRIAL: NCT05489016
Title: Prospective, Randomized, Double-blind, Placebo-controlled Clinical Study of Yuekang Huoxin Pill (Concentrated Pill) Intervening in the Prognosis of Patients With Coronary Heart Disease After Drug-Coated Balloon Implantation With Qi Deficiency and Blood Stasis Syndrome
Brief Title: HuoXin Pills Intervention on Patients With Coronary Heart Disease After Drug-Coated Balloon Implantation
Acronym: HAPPY-DCB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Fuwai Yunnan Cardiovascular Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Lihong Ma, Director of Department of Traditional Chinese Medicine, Principal Investigator, Clinical Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-1467
Record Dates: First submitted 2022-07-25; First posted 2022-08-05 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Coronary Heart Disease; Medicine, Chinese Traditional
Keywords: Coronary Heart Disease; Medicine, Chinese Traditional; Drug-coated balloon; Quantitative flow ratio
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yuekang Huoxin Pills (concentrated pills) (Experimental): 2 pills at a time, 3 times a day
  Interventions: Drug: Yuekang Huoxin Pills (concentrated pills)
- Yuekang Huoxin Pills (concentrated pills) simulant (Placebo Comparator): 2 pills at a time, 3 times a day
  Interventions: Drug: Yuekang Huoxin Pills (concentrated pills)simulant

INTERVENTIONS:
Drug: Yuekang Huoxin Pills (concentrated pills) — Huoxin Pill (concentrated pill) is composed of Radix Ginseng, Radix Aconiti Lateralis Preparata, Ganoderma, Flos Carthami, artificial Moschus, cultured calculus bovis in vitro, Fel Ursi, Margarita, Venenum Bufonis, and Borneolum Syntheticum. It has the effect of invigorating qi and promoting blood circulation. It has been marketed in China for more than 30 years. Clinical studies have shown that Huoxin Pill (concentrated pill) has significant clinical efficacy in improving the symptoms and prognosis of coronary heart disease and angina pectoris. Basic studies have also confirmed that Huoxin Pill (concentrated pill) can play a role in myocardial protection by dilating coronary arteries and promoting angiogenesis. It produced by Guangzhou yuekang biopharmaceuticals co., ltd.
  Arms: Yuekang Huoxin Pills (concentrated pills)
Drug: Yuekang Huoxin Pills (concentrated pills)simulant — Huoxin Pill (concentrated pill) simulant, a placebo-like simulation have no therapeutic effect. The shape, packaging and taste are the same as Huoxin Pill (concentrated pill), produced by Guangzhou yuekang biopharmaceuticals co., ltd.
  Arms: Yuekang Huoxin Pills (concentrated pills) simulant

SUMMARY:
This trial is a multi-center, randomized, double-blind, placebo, parallel controlled study. Objectively evaluates the curative effect of Huoxin Pills (concentrated pills) intervention on improving the prognosis of patients with coronary heart disease after drug-coated balloon implantation from a functional point of view. Huoxin Pill(concentrated pills), a traditional Chinese medicine, has been prescribed widely in the treatment of coronary heart disease, angina pectoris, and other diseases.440 patients were selected and followed up for one year. The quantitative blood flow score of the target vessel, late lumen loss, MACE incidence, and safety index were observed at 12 months.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is currently the main treatment for coronary heart disease. Drug-coated balloon (DCB) is an emerging interventional therapy technology. DCB can effectively reduce the incidence of vascular restenosis and cardiovascular composite event endpoints after PCI. However, the incidence of target lesion failure and major adverse cardiac event (MACE) of DCB in the treatment of primary coronary artery disease within one year after surgery can also reach more than 10%. Therefore, how to reduce vascular restenosis after DCB and other related cardiovascular composite endpoint events through the combination of DCB and drug therapy is a potential development direction of existing DCB therapy.

The research results of Chinese scholars have shown that the traditional Chinese medicine of replenishing qi and activating blood circulation can significantly reduce the restenosis rate after PCI, the recurrence rate of angina pectoris and the incidence of cardiovascular composite endpoint in three and six months after PCI.

It has significant clinical efficacy in improving the symptoms and prognosis of patients with coronary heart disease such as angina pectoris. In addition, basic research has further shown that Huoxin Pill (concentrated pill) can significantly reduce the degree and scope of myocardial ischemia and has the effects of dilating coronary artery and improving microcirculation.

Quantitative flow fraction (QFR) technology is the new method with the most sufficient clinical evidence in recent years, and can rapidly calculate the coronary stenosis-related lesions and severity of the diseased vessels in real time during the operation. Therefore, in this study, the QFR technology was used to evaluate the postoperative efficacy of DCB and the combination of Huoxin Pill (concentrated pill).

This trial is a multi-center, randomized, double-blind, placebo, parallel controlled study. Objectively evaluates the curative effect of Huoxin Pills (concentrated pills) intervention on improving the prognosis of patients with coronary heart disease after drug-coated balloon implantation from a functional point of view. Huoxin Pill(concentrated pills), a traditional Chinese medicine, has been prescribed widely in the treatment of coronary heart disease, angina pectoris, and other diseases.440 patients were selected and followed up for one year. The quantitative blood flow score of the target vessel, late lumen loss, MACE incidence, and safety index were observed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Patients who meet the diagnostic criteria of Western medicine for coronary heart disease, elective patients within two weeks after DCB surgery;
3. Voluntary selection of patients who undergo coronary angiography 12 months after surgery;
4. Meet the TCM criteria for syndrome differentiation of Qi deficiency and blood stasis (total score >= 8 points, and secondary symptoms >= 4 points);
5. The patients voluntarily participated in the trial and signed the informed consent.

Exclusion Criteria:

1. Severe arrhythmia, severe cardiopulmonary insufficiency and poorly controlled hypertension;
2. Patients with serious primary diseases such as severe liver and kidney damage, hematopoietic system, and mental illness;
3. Patients with heart valve disease, cardiomyopathy, congenital heart disease, aortic dissection or aortic aneurysm that need to be corrected by surgery or interventional therapy;
4. Those who have cerebrovascular events such as stroke and transient cerebral ischemia within 6 months;
5. Pregnant, planning pregnancy or lactating patients;
6. Allergic constitution and those who are allergic to known components of the research drug;
7. Those who are participating in other clinical trials or have participated in other drug clinical trials within one month;
8. Those who are judged by the investigator to be unsuitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
QFR | At the end of the 12-month follow-up
  quantitative flow fraction was measured by coronary angiography at 12-month follow-up. The AngioPlus system (Pulse Medical Imaging Technology, Shanghai Co., Ltd., Shanghai, China) is used for computation of QFR in this trial. n order to obtain accurate QFR measurement, analysts are required to follow the SOP (Standard Operation Procedure) for angiographic image acquisition.

SECONDARY OUTCOMES:
QFR change value | At the end of the 12-month follow-up
  quantitative flow fraction change value was measured by coronary angiography in 12-month Drug intervention. The AngioPlus system (Pulse Medical Imaging Technology, Shanghai Co., Ltd., Shanghai, China) is used for computation of QFR in this trial. n order to obtain accurate QFR measurement, analysts are required to follow the SOP (Standard Operation Procedure) for angiographic image acquisition.
Late Lumen Loss Late lume loss | At the end of the 12-month follow-up
  The software was used to automatically profile the artery by subtracting the minimum lumen diameter at the 12-month follow-up from the minimum lumen diameter immediately after coronary angiography within the drug-coating balloon.
incidence of main adverse cardiac events composite endpoints incidence of cardiovascular composite endpoints | At the end of the 12-month follow-up
  the occurrence of death, myocardial infarction and revascularization

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fuwai Hospital, China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes